CLINICAL TRIAL: NCT07369648
Title: Effects of Repetitive Transcranial Magnetic Stimulation Combined With Motor Rehabilitation on Motor and Functional Outcomes in Patients With Ischemic Stroke: A Randomized Sham-Controlled Trial
Brief Title: Repetitive Transcranial Magnetic Stimulation Combined With Motor Rehabilitation Improves Motor and Functional Outcomes After Ischemic Stroke
Acronym: rTMS-MOTOR
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Hanoi Medical University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: VN-2025-rTMS-MOTOR
Record Dates: First submitted 2026-01-18; First posted 2026-01-27 (Actual); Last update posted 2026-02-10 (Actual); Status verified 2025-12

CONDITIONS: Ischemic Stroke; Hemiplegia; Motor Function Impairment
Keywords: Repetitive Transcranial Magnetic Stimulation; rTMS; Motor Recovery; Post-Stroke Hemiplegia; Neurorehabilitation; Motor function
MeSH Terms: conditions — Ischemic Stroke; Hemiplegia

STUDY DESIGN:
Intervention Model Description: Participants are allocated into two parallel groups. The intervention group receives active repetitive transcranial magnetic stimulation combined with conventional motor rehabilitation, while the control group receives sham repetitive transcranial magnetic stimulation combined with the same conventional motor rehabilitation program. Participants are followed longitudinally, with outcome assessments conducted at baseline, immediately after completion of the intervention period, and at 3-month and 6-month follow-up assessments.
Who Masked: Participant, Outcomes Assessor
Masking Description: Participants are blinded using sham repetitive transcranial magnetic stimulation, in which the procedure, coil positioning, stimulation duration, and acoustic cues are identical to the active intervention, while the coil is positioned perpendicular to minimize cortical stimulation. Outcome assessors are blinded to group allocation and are not involved in participant recruitment, randomization, or intervention delivery. Assessments are conducted in a separate room and at different time points from the intervention sessions. In case of unintended unblinding, the assessor is replaced and the incident is documented.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Control Group (Placebo Comparator): Participants receive sham rTMS combined with the same standardized conventional motor rehabilitation program. Sham stimulation uses identical procedures, participant positioning, coil placement, session duration, and acoustic cues as active rTMS, but with the coil oriented perpendicular to the scalp to minimize effective cortical stimulation
  Interventions: Device: Sham repetitive transcranial magnetic stimulation; Other: Conventional motor rehabilitation
- Intervention Group (Experimental): Participants receive active low-frequency repetitive transcranial magnetic stimulation (rTMS) combined with standardized conventional motor rehabilitation targeting both upper and lower limb function. Active rTMS targets the primary motor cortex (M1) representations relevant to the upper limb (hand area) and lower limb (leg area), with stimulation parameters delivered according to the predefined protocol.
  Interventions: Device: Active repetitive transcranial magnetic stimulation; Other: Conventional motor rehabilitation

INTERVENTIONS:
Device: Active repetitive transcranial magnetic stimulation — Active rTMS is delivered at low frequency (1 Hz), 1200 pulses per session, 20 minutes per session, once daily, five days per week, for four consecutive weeks (20 sessions). rTMS is administered immediately prior to the daily conventional rehabilitation session.
  Upper limb target: Stimulation is applied to the M1 hand area using a figure-of-eight coil. The stimulation site is identified using standard localization methods (EEG 10-20 system landmarks and/or motor evoked potentials when available).
  Lower limb target: Stimulation is applied to the M1 leg area located near the cranial midline using a Hesed coil, with localization based on midline landmarks (near Cz) and/or motor evoked potentials from lower limb muscles when available.
  Stimulation intensity is set relative to the individual motor threshold.
  Arms: Intervention Group
Device: Sham repetitive transcranial magnetic stimulation — Sham rTMS is administered using the same procedures, participant positioning, coil placement, stimulation duration (20 minutes), and acoustic cues as the active stimulation protocol. To minimize effective cortical stimulation, the coil is oriented perpendicular to the scalp, producing minimal magnetic field penetration while preserving the characteristic clicking sound. Sham sessions follow the same schedule as active rTMS (once daily, five days per week, for four consecutive weeks; 20 sessions).
  Arms: Control Group
Other: Conventional motor rehabilitation — Participants receive standardized conventional motor rehabilitation for 60 minutes per day, five days per week, for four consecutive weeks. Each daily session includes three components: therapeutic exercise (approximately 20 minutes), physical therapy modalities (approximately 20 minutes), and occupational therapy/task-oriented functional training (approximately 20 minutes). The rehabilitation program is identical in content, intensity, and duration for both study arms.

SUMMARY:
Ischemic stroke is a leading cause of long-term motor disability, frequently resulting in hemiplegia and limitations in daily activities and quality of life. Motor rehabilitation is a fundamental component of post-stroke care across all stages of recovery; however, functional outcomes may vary, particularly in patients with persistent motor impairment.

Repetitive transcranial magnetic stimulation (rTMS) is a non-invasive brain stimulation technique that has been used as an adjunct to rehabilitation to modulate cortical excitability and potentially support motor recovery.

The purpose of this study is to evaluate the effects of low-frequency rTMS combined with conventional motor rehabilitation compared with sham rTMS combined with conventional motor rehabilitation in patients with first-ever ischemic stroke during the acute, subacute, and chronic stages. Motor function, balance, functional mobility, activities of daily living, and stroke-specific quality of life will be assessed at baseline, after the intervention, and at 3-month and 6-month follow-up.

DETAILED DESCRIPTION:
This study is a randomized, sham-controlled clinical trial designed to evaluate the outcomes of repetitive transcranial magnetic stimulation (rTMS) combined with motor rehabilitation in patients with first-ever ischemic stroke presenting with hemiplegia.Participants will be recruited during the acute (< 1 month), subacute (1-6 months), and chronic (> 6 months) stages after stroke onset.

Eligible participants will be allocated into two groups: a control group and an intervention group. Both groups will receive standardized conventional motor rehabilitation targeting upper and lower limb motor function, balance, and functional mobility.

In the intervention group, participants will receive low-frequency rTMS in addition to conventional motor rehabilitation. rTMS will be delivered at a frequency of 1 Hz, once daily, five days per week, for a total of 20 sessions. For upper limb rehabilitation, stimulation will be applied to the primary motor cortex (M1) corresponding to the hand area of the contralesional hemisphere using a figure-of-eight coil. For lower limb rehabilitation, stimulation will target the leg area of M1 located in the medial interhemispheric region using a Hesed coil. Stimulation intensity will be set relative to each participant's motor threshold, and rTMS sessions will be administered immediately prior to motor rehabilitation.

In the control group, participants will receive sham rTMS combined with the same conventional motor rehabilitation program. Sham stimulation will be performed using identical procedures, participant positioning, coil placement, stimulation duration, and acoustic output as the active rTMS condition. To minimize cortical stimulation, the coil will be positioned perpendicular to the scalp, producing minimal magnetic field penetration while maintaining the characteristic clicking sound of the device.

To ensure blinding, participants will not be informed of their group allocation, and they will be instructed not to disclose any information related to the intervention they received prior to outcome assessments. Outcome assessors will be blinded to group assignment.

Outcome measures will be assessed at baseline, immediately after completion of the intervention, and at 3-month and 6-month follow-up to evaluate motor recovery, balance, functional mobility, activities of daily living, and stroke-specific quality of life.

ELIGIBILITY:
Inclusion Criteria:

* Aged 18 to 80 years.
* Diagnosed with a first-ever ischemic stroke, confirmed by neuroimaging.
* Presence of unilateral hemiparesis attributable to the first-ever ischemic stroke.
* Time since stroke onset:

  * Acute stage: < 1 month after stroke onset
  * Subacute stage: 1 to 6 months after stroke onset
  * Chronic stage: > 6 months after stroke onset
* Moderate neurological impairment, defined as a baseline NIHSS score between 5 and 14.
* Cognitive ability sufficient to understand and follow instructions, indicated by a baseline MMSE score ≥ 20.
* Medically stable and able to participate in a structured motor rehabilitation program.
* Provided written informed consent prior to study enrollment.
* NIHSS and MMSE scores are assessed at baseline only to characterize neurological severity and cognitive status at study entry

Exclusion Criteria:

* Motor impairment caused by conditions other than ischemic stroke, such as musculoskeletal disorders, traumatic brain injury, Parkinson's disease, encephalitis, or other neurological conditions.
* Contraindications to repetitive transcranial magnetic stimulation, including but not limited to intracranial metallic implants, implanted electronic medical devices (e.g., pacemaker), cochlear implants, known bleeding disorders, pregnancy, history of epilepsy or seizure disorders, severe cardiac disease, severe psychiatric or neurological disorders interfering with participation, or active skin conditions at the stimulation site.
* History of epilepsy or seizure disorders.
* Recurrent stroke occurring during the intervention period.
* Refusal to participate, withdrawal of informed consent, or non-adherence to the intervention protocol.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 66 (Estimated)
Dates: Start 2026-02 (Estimated); Primary Completion 2027-06 (Estimated); Study Completion 2028-12 (Estimated)

PRIMARY OUTCOMES:
Change in upper limb motor function assessed by the Fugl-Meyer Assessment for Upper Extremity (FMA-UL) | Baseline, immediately after the 4-week intervention period, and at 3-month and 6-month follow-up
  The Fugl-Meyer Assessment for Upper Extremity (FMA-UL) is a validated scale for evaluating motor impairment of the upper limb after stroke. Scores range from 0 to 66, with higher scores indicating better motor function.

SECONDARY OUTCOMES:
Change in manual dexterity assessed by the Box and Block Test (BBT) | Baseline, immediately after the 4-week intervention period, and at 3-month and 6-month follow-up
  The Box and Block Test assesses gross manual dexterity by counting the number of blocks transferred within 60 seconds
Change in functional mobility assessed by the Timed Up and Go test (TUG) | Baseline, immediately after the 4-week intervention period, and at 3-month and 6-month follow-up
  The Timed Up and Go test measures functional mobility and balance by recording the time required to stand up, walk, turn, and sit down
Change in balance performance assessed by the Berg Balance Scale (BBS) | Baseline, immediately after the 4-week intervention period, and at 3-month and 6-month follow-up
  The Berg Balance Scale evaluates static and dynamic balance abilities, with scores ranging from 0 to 56
Change in activities of daily living assessed by the modified Barthel Index (mBI) | Baseline, immediately after the 4-week intervention period, and at 3-month and 6-month follow-up
  The modified Barthel Index measures independence in activities of daily living, with higher scores indicating greater functional independence
Change in quality of life assessed by the Stroke-Specific Quality of Life Scale (SS-QoL) | Baseline, immediately after the 4-week intervention period, and at 3-month and 6-month follow-up
  The Stroke-Specific Quality of Life Scale assesses health-related quality of life across multiple domains in stroke survivors

CONTACTS AND LOCATIONS:
Overall Officials: Loan Phan Thi Kieu, MD, MSc, Principal Investigator — Hanoi Medical University, Hanoi, Vietnam

IPD SHARING:
Plan to Share IPD: Yes
De-identified individual participant data, including demographic information, baseline characteristics, intervention allocation, and outcome measures collected during the study, will be shared. All shared data will be fully anonymized and will not contain any information that could identify individual participants.
Supporting Information: Study Protocol, SAP
Time Frame: Beginning 6 months after publication of the primary results and ending 5 years thereafter.
Access Criteria: Data will be shared upon reasonable request from qualified researchers. Requests will be reviewed by the study investigators and require approval of a research proposal and a data use agreement.